CLINICAL TRIAL: NCT05925972
Title: Effects of Ultrasonography-Guided Plan Blocks (ESP&OSTAP) on Perioperative Analgesia in Laparoscopic Hysterectomies
Brief Title: Analgesic Efficacy of Plan Blocks in Laparoscopic Hysterectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Nazan KOCAOGLU, MD, Assistant professor, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DT/2022-04-01
Record Dates: First submitted 2023-06-06; First posted 2023-06-29 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup ESP (Active Comparator): The group to which erector spina plane block will be applied
  Interventions: Procedure: Plane block
- Grup OSTAP (Active Comparator): The group to which oblique subcostal transversus abdominis plane block will be applied
  Interventions: Procedure: Plane block

INTERVENTIONS:
Procedure: Plane block — Plane block application in laparoscopic hysterectomies

SUMMARY:
Hysterectomy is the most common major intervention in gynecology after cesarean section. Indications include myoma uteri, abnormal uterine bleeding, cervical intraepithelial neoplasia, chronic pelvic pain, uterine uteri, operated breast cancer, and endometrial hyperplasia. Today, hysterectomy can be performed abdominally, vaginally and laparoscopically.¹ Laparoscopic hysterectomy (LH) has several advantages and disadvantages compared to other forms of hysterectomy. Shorter recovery time, less wound infection, shorter hospital stay, and less need for postoperative analgesia can be counted among the advantages. The prolongation of the operation time and the increased risk of urinary complications are disadvantages.² Postoperative pain management can be done with different methods depending on the location of the surgical field, the type of surgical procedure, the patient's need for analgesia, and patient preference. These methods include oral, intravenous or intramuscular medication and nerve blocks. In order to minimize the side effects of opioids used in analgesic therapy such as respiratory depression, nausea-vomiting, lethargy, constipation and itching, and to increase the analgesic effect, the "balanced analgesia" method is used.⁴ With this method, opioids, non-opioid analgesics or peripheral nerve-field blocks side effects are minimized and optimum analgesia is provided.

Transversus abdominis plane (TAP) block, which is one of the abdominal field blocks, was first described by Rafi in 2001.⁶ Hebbard et al. stated in 2007 that ultrasonography (USG)-guided TAP block can be applied more effectively and safely.⁷ This block can be applied more effectively and safely.⁷ This block is antero-lateral, posterior, and oblique It can be done subcostal with three different approaches. TAP block has been shown to reduce postoperative pain after hysterectomy, cesarean section, and colorectal surgery.⁸ Erector spina plane (ESP) block was first described by Forero et al. in 2016 on a patient with chronic neuropathic pain.⁹ The basic technique is performed paraspinally under USG guidance. It is used for postoperative analgesia in breast, thoracic surgeries, hernia repair, dorsal colon, abdomen and hip surgery.

In this study, it is aimed to compare the effects of USG-guided ESP block and OSTAP block applications on perioperative pain control in total laparoscopic hysterectomy operations.

DETAILED DESCRIPTION:
MATERIAL AND METHOD Patients between the ages of 18-65, ASA I-II, BMI ≤30 kg/m2 who will undergo elective surgery under general anesthesia, with voluntary consent will be included in the study. Patients with local anesthetic allergy, coagulopathy, infection at the block application site, and mental deficiency and for whom the surgical plan has been changed (complicated/open surgery) will be excluded from the study.

Patients included in the study will be informed about patient-controlled analgesia (PCA) and numerical rating scale (NRS: Numeric Rating Scale) for the assessment of pain severity before the operation. Demographic data of the patients will be recorded.

Anesthesia Application:

After the intravenous (IV) route is provided with a 20 G cannula in the preoperative preparation room, 10 mL/kg of balanced crystalloid fluid infusion will be started. 0.03 mg/kg midazolam will be administered for premedication. Standard monitoring (ECG, heart rate, non-invasive blood pressure, SPO2, temperature) and neuromuscular monitoring will be applied to all patients. The input value of these parameters will be saved before induction. Records will be taken at 5-minute intervals until the end of the operation. For induction of anesthesia, 2 mg/kg propofol, 1μg/kg remifentanil will be administered as an IV bolus within 60 seconds. Analgesia maintenance will be provided with 0.05-0.25 μg/kg/min remifentanil infusion. Muscle relaxation will be provided with IV 0.6 mg/kg rocuronium. He will be intubated orotracheally when his train of four rate (TOFR) response is zero. (In case of neuromuscular blocker requirement, IV 0.01 mg/kg rocuronium will be additionally administered.) Anesthesia is maintained with 0.5 L/min fresh gas flow, oxygen concentration with inspiratory oxygen level between 40-45, minimum alveolar concentration (MAC) with 0.9-1.1 with sevoflurane. will be applied. Mechanical ventilation will be performed with Volume AutoFlow mod (V-AF) with ETCO2 between 35-40 mmHg.

Patients will be randomly divided into two groups after induction. Group ESP (I): The group to which Erector Spina Plan Block (ESP) will be administered Group OSTAP (II): The group to which Oblique Subcostal Transversus Abdominis Plan Block (OSTAP) will be applied In the study, anesthesia induction and plan blocks will be performed by the same anesthesiologist. Intraoperative and postoperative data recording and patient evaluation will be done by two separate anesthesiologists.

ESP Block Application:

In the lateral decubitus position after induction, in accordance with the rules of asepsis-antisepsis, USG (Sonosite M-Turbo) machine, linear 6-13 mHz probe will be placed approximately 3 cm lateral to the T9 spinous process in the sagittal plane and with an in-plane approach, the hyperechoic shadow of the transverse process and the erector spina muscle ( Once the ESM) has been identified, a 22 G, 80 mm Stimuplex® Ultra 360® (B.Braun, Melsungen, Germany) needle will be inserted in the cephalocaudal direction to gently contact the T9 spinous process over the erector spinae. After negative pressure aspiration between the transverse process and ECM, 1-2 mL of local anesthetic will be injected, and after cephalocaudal spread is observed, a total of 20 mL of 0.25 mg/mL bupivacaine will be given by intermittent aspiration every 4-5 mL. The same procedure will be applied to the other side.

OSTAP Block Application:

After the induction, in the supine position, in accordance with the rules of asepsis-antisepsis, the USG (Sonosite M-Turbo) machine will be placed on the anterior axillary line, the linear 6-13 mHz probe will be placed on the subcostal lower edge between the xiphoid and the anterosuperior iliac process, and the rectus abdominis and transversus abdominis muscles will be visualized. Then, 22 G, 80 mm Stimuplex®Ultra 360® (B.Braun, Melsungen, Germany) needle is directed in-plane from 2-3 cm medial of the rectus abdominis muscle, negative pressure aspiration between the transversus abdominis and rectus abdominis muscles is applied 1-2 mL of local anesthetic will be injected. After local anesthetic spread is observed, a total of 20 mL of 0.25 mg/mL bupivacaine will be given by intermittent aspiration every 4-5 mL. The same procedure will be applied to the other side.

Surgical incision will be made 15 minutes after block applications. Patients will undergo standard surgical procedures. The patients will be operated in the 45⁰ trendelenburg position and the pneumoperitoneum pressure is 10-12 mmHg. In case of (±) 15% change in the hemodynamic parameters of the patient compared to the initial values, the remifentanil infusion dose will be increased or decreased at the specified intervals and the amount consumed intraoperatively at the end of the operation will be recorded. It will be defined as hypotension when the systolic arterial pressure decreases by 30% from the baseline value. In the treatment, 250 mL of 0.9% NaCl will be rapidly infused first. If there is no response, 10 mg of ephedrine will be given IV. When bradycardia occurs (heart rate <50 beats/min) IV 0.5 mg of atropine will be administered. The time from the skin incision to the end of the surgical procedure will be recorded as "Operation Time".

Sevoflurane flow and remifentanil infusion will be terminated 15 minutes before the end of the operation. Patients will be administered 50 mg dexketoprofen trometamol IV and 1 g paracetamol IV infusion. At the end of the operation, the fresh gas flow will be increased to 8 L/min. To end the neuromuscular blockade, 4 mg/kg of sugammadex will be administered IV. When the TOFR is 0.9, he will be extubated and transferred to the postoperative recovery unit (PACU). The time between termination of sevoflurane flow and extubation will be recorded as "Extubation time", and the time between anesthesia induction and extubation will be recorded as "Anesthesia Time".

Patient-controlled analgesia (PCA) and morphine infusion will be administered to both groups of patients in the PACU.

Morphine protocol: It will be prepared as 1 mg/mL with 5 mL Morphine Sulphate (50mg) + 45 mL physiological saline. It will be administered as an intermittent bolus of 1 mg, without basal infusion, with a 20-minute lock-in time.

Postoperative pain intensity, sedation level and nausea-vomiting score of the patients at rest and movement status will be evaluated at 0, 2, 4, 6, 12 and 24 hours by an anesthesiologist who is not familiar with the study groups.

The severity of pain will be evaluated with NRS at rest and in motion (0: No pain 1 2 3 4 5 6 7 8 9 10: Unbearable pain) If NRS≥4, dexketoprofen trometamol 50 mg IV will be administered as a rescue analgesic.

The Observer's Assessment of the Alertness/Sedation (OAA/S) will be used to monitor the sedation level of the patient.

Nausea will be measured with 4 categorical scoring systems (No nausea: 0, Mild: 1, Moderate: 2, Severe: 3) For the treatment of nausea-vomiting, 4mg ondansetron will be administered IV. Patients with a modified Aldrete score ≥9 will be discharged to the ward. The time elapsed between the patient's admission to the PACU and discharge to the service will be recorded as "Recovery Time".

ELIGIBILITY:
Inclusion Criteria:

Between 18-65 years laparoscopic hysterectomy under general anesthesia ASA I-II BMI ≤30 kg/m2

Exclusion Criteria:

local anesthetic allergy coagulopathy infection at the block application site mental deficiency the surgical plan has been changed (complicated/open surgery)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-12-14 (Actual)

PRIMARY OUTCOMES:
Plane blocks | Intraoperative and postoperative first 24 hours
  Analgesic efficacy between ESP and OSTAP blocks will be evaluated by Numeric Rating Scale. Intraoperative and postoperative opioid consumption will be compared.

SECONDARY OUTCOMES:
Nausea | Intraoperative and postoperative first 24 hours
  Nausea, vomiting and other side effects will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Nazan Kocaoglu, Principal Investigator — Balikesir University Medical Faculty
Locations (2):
- Turkey (Türkiye) (2):
  - Balikesir University, Balıkesir
  - Medical faculty, Balıkesir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Result] Abdallah FW, Chan VW, Brull R. Transversus abdominis plane block: a systematic review. Reg Anesth Pain Med. 2012 Mar-Apr;37(2):193-209. doi: 10.1097/AAP.0b013e3182429531. PMID 22286518

DOCUMENTS (1):
  • Study Protocol (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT05925972/Prot_000.pdf